CLINICAL TRIAL: NCT04693572
Title: Anesthetic Considerations for Repeat Cesarean Section - a Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Jacob Weinstein, MD MSc, Clinical Fellow, Shaare Zedek Medical Center
Other Study IDs: 0415-20-SZMC
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Anesthesia; Pregnancy, High Risk; Pregnancy Related
Keywords: Caesarian Section; Repeated Caesarian Section; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parturients undergoing repeated caesarean sectiona

SUMMARY:
The purpose of this study is to examine the anesthetic considerations and outcomes during repeated caesarean section and to compare such considerations in low-order vs high-order repeated caesarean sections.

DETAILED DESCRIPTION:
Data concerning anesthetic considerations and outcomes will be gathered from the electronic medical records of all parturients undergoing repeated caesarean sections in our medical center. the collected data will be stored anonymously.

Different aspects of anesthetic considerations and outcomes will be compared and subjected to analysis.

ELIGIBILITY:
Inclusion Criteria:

* Parturients undergoing repeated caesarean section.

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parturients undergoing repeated caesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of sections performed under general anesthesia | 1 day
Percentage of in-surgery conversion from regional to general anesthesia | 1 day

IPD SHARING:
Plan to Share IPD: Undecided